CLINICAL TRIAL: NCT07350525
Title: CASTomize 4D Printed Cast Versus Fibreglass Casts for Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, YAM GUI JIE MICHAEL, Dr, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/00073
Record Dates: First submitted 2025-12-31; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Standard of care cast
  Interventions: Other: Control
- Intervention (Experimental): Castomize cast arm
  Interventions: Device: Castomize cast

INTERVENTIONS:
Device: Castomize cast — 4D castomize cast for distal radius fracture immobilisation
  Arms: Intervention
Other: Control — Standard of care casting
  Arms: Control

SUMMARY:
This study is a randomised control trial comparing Castomize 4D printed cast versus conventional fibreglass casts in isolated conservatively treated distal radius fractures. The primary outcome measure is fracture reduction. Secondary outcome measures include patient reported outcome measures such as the Adult Rated Cast Evaluation Questionnaire (ARCEQ), comfort of the cast, quality of life assessed with the EQ-5D-5L questionnaire, cost-effectiveness and adverse events occurrence. In total, 30 patients will be included and followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 21 years
* Distal radius fracture for conservative treatment within 3 weeks of initial injury

Exclusion Criteria:

* Concomitant injuries to the ipsilateral extremity, interfering with the treatment of the DRF (Example: concomitant elbow fracture that requires further immobilisation with a above elbow cast)
* Inability to complete study forms due to any cognitive, mental issues.
* Pregnant women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-01-14 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
Fracture reduction | 3 months
  Fracture alignment is determined by length rotation and angulation in clinically acceptable values as determined by surgical team

SECONDARY OUTCOMES:
comfort, pain, itch | 6 months
  Quantitative Likert scoring for comfort, pain, itch as well as qualitative feedback on cast application and comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT07350525/Prot_SAP_000.pdf